CLINICAL TRIAL: NCT03017690
Title: Lanreotide and Octreotide LAR for Patients With Advanced Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs): An Observational Time and Motion Analysis
Brief Title: Lanreotide and Octreotide Long Acting Release (LAR) for Patients With Advanced Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs)
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-US-52030-358
Record Dates: First submitted 2016-12-30; First posted 2017-01-11 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lanreotide group (Somatuline Depot®)
- octreotide LAR group (Sandostatin LAR®)

SUMMARY:
An observational time and motion study in a clinical oncology setting is utilized in order to measure and compare product attributes and overall product efficiency between lanreotide and octreotide LAR.

ELIGIBILITY:
Inclusion Criteria:

* Men and women must be 18 years of age or older
* A current diagnosis of advanced, unresectable GEP-NET
* Provided written informed consent to participate in the study
* Currently receiving lanreotide or octreotide LAR and has received at least one prior injection of current somatostatin analogues (SSA).

Exclusion Criteria:

* Receiving treatment with lanreotide or octreotide LAR as part of a clinical trial
* Scheduled to receive a dose of lanreotide or octreotide LAR that would necessitate more than 1 injection on the same day
* Scheduled to receive any other treatment in the infusion center/room on the same day and as part of the same appointment
* Known hypersensitivity to somatostatin analogues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited through US institutions/clinics that commonly treat neuroendocrine tumor patients.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
The total time for product preparation and administration | Day 1
  Total drug delivery time

SECONDARY OUTCOMES:
Total patient wait time for administration | Day 1
  For the purposes of this study, "total patient wait time" refers to the time the patient checks in at the infusion room until completion of drug administration and discharge of the patient from the infusion room.
Number of clogging episodes | Day 1
  The number of clogging episodes for lanreotide and octreotide LAR will be recorded and compared.
Healthcare resource utilization | Day 1
  The materials used for the preparation of lanreotide and octreotide LAR will be recorded and compared.
Pharmacist and/or nurse satisfaction and product preference | Day 1 and at the end of the study (approximately 3 months)
  Assessed by pharmacist and/or nurse completing questionnaire
Patient satisfaction | Day 1
  Assessed by patient completing questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (5):
- United States (5):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - National Translational Research Group, East Setauket, New York
  - Oncology Specialists of Charlotte, Charlotte, North Carolina

REFERENCES:
- [Derived] Ryan P, McBride A, Ray D, Pulgar S, Ramirez RA, Elquza E, Favaro JP, Dranitsaris G. Lanreotide vs octreotide LAR for patients with advanced gastroenteropancreatic neuroendocrine tumors: An observational time and motion analysis. J Oncol Pharm Pract. 2019 Sep;25(6):1425-1433. doi: 10.1177/1078155219839458. Epub 2019 Mar 29. PMID 30924737